CLINICAL TRIAL: NCT01544881
Title: A Phase 1, Single-center, Open-label, Randomized, Crossover Design Clinical Study in Subjects With Type 1 Diabetes Comparing Insulin Exposure & Response Following Inhalation of Technosphere Insulin Inhalation Powder Using the Gen2C Inhaler Vs Subcutaneous Rapid-Acting Analog
Brief Title: Comparison of Technosphere Insulin Inhalation Powder & Subcutaneous Rapid-Acting Analog in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MKC-TI-177
Record Dates: First submitted 2012-02-23; First posted 2012-03-06 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Pharmacokinetics; Pharmacodynamics; Hyperglycemia; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TI Inhalation Powder (Experimental): Technosphere Insulin Inhalation Powder using the Gen2C inhaler
  Interventions: Drug: Technosphere Insulin Inhalation Powder
- RAA (Active Comparator): Rapid Acting Analog
  Interventions: Drug: Rapid Acting Analog

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder — Inhalation Powder using the Gen2C inhaler
  Other Names: TI
  Arms: TI Inhalation Powder
Drug: Rapid Acting Analog — Subcutaneous Injection
  Other Names: RAA
  Arms: RAA

SUMMARY:
This is an Open-label, randomized study in Type 1 diabetics looking at exposure and response (PK/PD) of TI using GEN2C Inhaler versus rapid acting analog.

DETAILED DESCRIPTION:
Subjects with Type 1 diabetes will be randomized to either one dose of TI inhaled using the Gen2C device, or one dose of subcutaneously injected Rapid Acting Analog (RAA) and crossed over.

Crossover Sequences:

Sequence #1: Period 1 - one 20 U cartridge of TI; Period 2 - 8 U of RAA

Sequence #2: Period 1 - 8 U RAA; Period 2 - one 20 U cartridge of TI

An euglycemic clamp procedure will be performed at each dosing visit. The purpose of this study is to characterize the pharmacokinetics (PK) of the one dose of TI Inhalation Powder using the Gen2C inhaler as compared to one dose of subcutaneous RAA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 60 years
* One of more daily sc insulin injections of any insulin type or insulin pump use
* Body mass index (BMI) = 30 kg/m2
* Pulmonary function tests (PFTs) conducted at Visit 1:

  * FEV1 ≥ 80% of the Third National Health and Nutrition Examination Survey (NHANES III) predicted
  * FVC ≥ 80% of the Third National Health and Nutrition Examination Survey (NHANES III) predicted
* Diagnosis of type 1 diabetes for at least 12 months
* Good venous access for blood draws
* Written informed consent provided
* No smoking in the previous 6 months (including cigarette, cigars, pipes) and negative urine cotinine testing (<100 ng/mL)
* C-peptide < 0.3 ng/mL
* Hemoglobin A1c (HbA1c) = 10.0%

Exclusion Criteria:

* Total daily insulin requirement of = 1.4 U/kg body weight
* Serum creatinine = 2.0 mg/dL in men and > 1.8 mg/dL in women
* Blood donation of 500 mL within the previous 56 days
* Current treatment with pramlintide acetate or exenatide
* Unstable diabetes control and evidence of severe complications of diabetes (ie, autonomic neuropathy)
* History of chronic obstructive pulmonary disease (COPD) or asthma, or any other clinically important pulmonary disease confirmed by pulmonary function testing or radiologic findings
* Upper respiratory tract infection within 8 weeks before screening
* History of coronary artery disease, peripheral vascular disease, or congestive heart failure
* Allergy to study drug, food, or other study material (eg, peanuts, soy products)
* Clinically significant active or chronic illness
* History of drug or alcohol abuse
* Positive urine drug screen
* Clinically significant screening ECG, physical examination, laboratory test, or vital sign abnormality
* Exposure to any other investigational drug or device within 30 days before treatment or within 90 days before treatment for drugs known to modify glucose metabolism (except metformin)
* History of malignancy within the 5 years before screening (other than basal cell carcinoma)
* History of human immunodeficiency virus (HIV) infection or hepatitis B or C
* Women who are pregnant, lactating, or planning to become pregnant during the clinical study period
* Women of childbearing potential (defined as premenopausal and not surgically sterilized or postmenopausal for fewer than 2 years) not practicing adequate birth control. Adequate birth control is defined as using oral, percutaneous, or transdermal contraceptives; condoms and diaphragms (double barrier) with a spermicide; or intrauterine devices. Postmenopausal for the purposes of this clinical study includes experiencing amenorrhea for 2 or more years or being surgically sterile
* Inability, in the opinion of the PI or a designee, to adequately inhale TI Inhalation Powder
* Any subject who, in the opinion of the PI or a designee, appears to not be qualified for this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
PK measures for TI Inhalation Powder (20U) as measured by area under the concentration-time curve (AUC 0-360) - timepoints: 0, 3, 6, 9, 12, 15, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 240, 300 and 360 minutes post-TI dosing | Crossover 1 time within 3 - 10 days
PK measures for RAA (8U) as measured by area under the concentration-time curve (AUC 0-360) - timepoints 0, 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, 300 and 360 minutes post-RAA dosing | Crossover 1 time within 3 - 10 days

SECONDARY OUTCOMES:
Safety variables including adverse events (AEs), clinical laboratory tests, vital signs and physical examinations | Crossover 1 time within 3 - 10 days
Area under serum glucose infusion rate (GIR AUC 0-360) for TI Inhalation Powder (20U) as measured by: GIR AUC 0-360 timepoints: 0, 3, 6, 9, 12, 15, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 240, 300 and 360 minutes post-TI dosing | Crossover 1 time within 3 - 10 days
Area under serum glucose infusion rate (GIR AUC 0-360) for RAA (8U) as measured by: GIR AUC 0-360 timepoints: 0, 5, 10, 15, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, 300 and 360 minutes post-RAA dosing | Crossover 1 time within 3 - 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Mannkind Corporation
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States